CLINICAL TRIAL: NCT06955312
Title: The Effect of Paint-by-Numbers Activity on Stress and Prenatal Attachment in High-Risk Pregnancies
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erzurum Technical University (Other)
Collaborators: Scientific Research Projects Coordination Unit (Ambiguous)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 22
Record Dates: First submitted 2025-02-27; First posted 2025-05-02 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-02

CONDITIONS: High-Risk Pregnancies
Keywords: High-risk pregnancy; Prenatal attachment; Stress management; Paint-by-numbers activity; Randomized controlled trial

STUDY DESIGN:
Intervention Model Description: The G*Power program (version 3.1.9.3) was used to calculate the sample size, and Cohen's standard effect size was considered for determining the sample size. According to Cohen, an effect size of 0.20 is classified as "small," 0.50 as "medium," and 0.80 as "large." In this study, Cohen's effect size was assumed to be 0.80 to determine the minimum required sample size. Based on this effect size, the Type I error was set at 0.05, and the power of the test was 0.80 (α = 0.05, 1-β = 0.80, effect size = 0.80). As a result, the required sample size for the study was determined to be 52 participants (n = 26 per group) for an equal distribution between groups. Considering potential participant dropout, the final sample size was determined to be 60 participants (n = 30 per group).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Experimental): Experimental group pregnant women will be asked to paint with numbers of 40x50cm canvases containing mother and baby. Pregnant women will be asked to paint the table according to their own wishes and finish them in about 5 days.
  Interventions: Behavioral: Experimental
- Group B (No Intervention): This group will take routine care applications

INTERVENTIONS:
Behavioral: Experimental — Description: After collecting the pre-test data, pregnant women in the experimental group will be informed about the paint-by-numbers activity, and the materials to be used will be introduced. Participants in the experimental group will be asked to choose one of the 40x50 cm paintings. They will then be instructed to complete the painting. Pregnant women will be asked to paint the selected canvas at their convenience over approximately five days. Once the paint-by-numbers activity is completed, participants will be asked to fill out the post-test questionnaires, and final data from the experimental group will be collected, marking the end of the data collection process. After data collection, participants will be gifted their completed paintings, which they can hang in their children's rooms.
  Arms: Group A

SUMMARY:
Pregnancy, a physiological state, is defined both as a turning point and a developmental crisis . Pregnancy directly affects maternal and child health, and in cases of complications, it can lead to morbidity and mortality, particularly in developing countries . According to data from the World Health Organization (WHO), approximately 830 women worldwide die daily due to preventable pregnancy- and childbirth-related causes, with 99% of all maternal deaths occurring in developing countries, including Turkey (https://www.who.int/news-room/fact-sheets/detail/maternal-mortality).

In Turkey, the 2005 National Maternal Mortality Study reported a maternal mortality rate of 28.5 per 100,000 live births. This study revealed that 49.3% of pregnancy-related deaths and 61.6% of maternal deaths were due to preventable causes Hemorrhage, infection, and preeclampsia/eclampsia are among the leading causes of maternal mortality both in Turkey and globally . This significant issue is included in the Sustainable Development Goals (2016-2030) as a target to reduce global maternal mortality

High-risk pregnancy refers to conditions where maternal, fetal, or neonatal health is partially or entirely at risk . According to the 2013 Turkey Demographic and Health Survey (TNSA), 63% of pregnant women aged 18-34 in Turkey fall into at least one risk category. High-risk pregnancies are associated with various physiological and psychological challenges, negatively impacting maternal, infant, and family health . In addition to posing life-threatening risks, high-risk pregnancies represent a crisis related to fertility . When a pregnancy is high-risk, emotional distress increases due to maternal or fetal complications . Compared to low-risk pregnancies, high-risk pregnant women experience significantly higher stress regarding their own and their baby's health .

Stressors experienced by high-risk pregnant women include receiving a high-risk pregnancy diagnosis, unplanned pregnancy, pregnancy complications, fetal abnormalities, childbirth fears, adolescent pregnancies, marital issues, lack of social support, economic concerns, postpartum problems, and hospitalization . Perceived stress during pregnancy is highly significant for pregnancy outcomes . Pregnancy-related stress has been characterized as a stronger form of stress than general stress due to its ability to trigger heightened physiological arousal . This can have adverse effects, increasing maternal and fetal morbidity and mortality risks . Stress may elevate oxytocin and prostaglandin hormone levels while reducing beta-endorphin and progesterone levels, leading to birth complications or adverse birth outcomes .

Stress during pregnancy has been associated with negative birth outcomes, including preterm labor, spontaneous abortion, neonatal malformations, and growth retardation . Additionally, stress can negatively impact parental attachment to the fetus and newborn . There is a bidirectional relationship between attachment and a woman's psychosocial well-being. Prenatal attachment is influenced by the mother's psychosocial state, and a lack of attachment can negatively affect her mental well-being. Literature suggests a link between prenatal attachment and long-term maternal depression . A study highlighting the potential adverse effects of stress on prenatal attachment in high-risk pregnancies emphasized the importance of supporting prenatal attachment to prevent postpartum issues such as anxiety and depression .

DETAILED DESCRIPTION:
Stress, which has adverse effects even in the postpartum period, is among the modifiable risk factors in high-risk pregnancies. A study published in The Lancet on maternal health reported that at least 40 million women worldwide experience long-term health problems due to childbirth. The study highlighted persistent issues such as anxiety (9-24%), depression (11-17%), and tokophobia (6-15%) months or even years after delivery (Vogel et al., 2024). Many of these conditions are thought to stem from poorly managed stress. A study in Nepal identified stressful life events as contributing factors to postpartum depression symptoms .

Negative pregnancy outcomes not only affect maternal and infant health but also place a significant economic burden on countries. For instance, in the United States, the annual costs associated with preterm birth-including medical care, parental work loss, and specialized education-are estimated at $26 billion. Literature underscores that effective care during pregnancy and childbirth is a crucial preventive factor in identifying risks and preventing complications that could lead to long-term health issues. The International Council of Nurses (ICN) states that nurses play a vital role in educating individuals about what they need to maintain good health.

Hospitalization can create stress for high-risk pregnant women, highlighting the importance of introducing activities that help manage stress during this period. A review of the literature revealed no randomized controlled studies examining the effects of a paint-by-numbers activity on perceived stress and prenatal attachment in hospitalized high-risk pregnant women. This study aims to investigate the effects of a paint-by-numbers activity on stress and prenatal attachment among high-risk pregnant women receiving inpatient care at Erzurum City Hospital. It is anticipated that this study will contribute to reducing stress and enhancing prenatal attachment among women with high-risk pregnancies. Additionally, it is expected to raise awareness among healthcare providers, particularly nurses, about incorporating such activities into their care practices.

ELIGIBILITY:
Inclusion Criteria:

* Having a high-risk pregnancy
* Being at or beyond the 20th week of pregnancy
* Being hospitalized for at least 4 days for high-risk pregnancy monitoring
* Being open to communication and collaboration
* Being literate in Turkish
* Being over 18 years of age
* Volunteering to participate in the study

Exclusion Criteria:

* Being under 18 years of age

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — High-risk pregnancy
Enrollment: 60 (Estimated)
Dates: Start 2025-05-15 (Estimated); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-09-10 (Estimated)

PRIMARY OUTCOMES:
Perceived Stress Level | 10-15 Minutes
  Measured using a validated stress scale (Perceived Stress Scale in High-Risk Pregnancies Based on the Neuman Systems Model (NSM-HRPS). The lowest possible score from NSMt-RGASÖ is 34 and the highest is 170. While the sum of the scores in the sub-dimensions in NSMt-RGASÖ constitutes the stress score in that life area, the sum of the scores of all the items constitutes the total scale score. A high score from the overall scale and the sub-dimensions indicates that the perceived stress in the relevant life area and in general is high.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe METİN, Assistant Professor (Dr.), Study Director — Erzurum Technical University Faculty of Health Sciences

IPD SHARING:
Plan to Share IPD: No
Confidentiality and Ethical Considerations:
  The study involves sensitive health-related data from high-risk pregnant women, making it essential to protect participant privacy.
  Ethical guidelines and data protection regulations (e.g., GDPR, HIPAA) restrict the sharing of personally identifiable information.
  Institutional and Legal Restrictions:
  The data is collected under specific institutional and national regulations that may limit external access.
  Institutional Review Board (IRB) or Ethics Committee approval may be required for any data-sharing requests.
  Data Security and Misuse Prevention:
  To prevent misinterpretation or misuse, raw data will not be publicly available.
  Only aggregated results and summary findings will be shared in publications or upon request.
  Limited Resources for Data Management:
  Providing external access requires additional resources for data anonymization, secure storage, and compliance monitoring.
  The research team may not have the capacity to manage extern

REFERENCES:
- [Background] Vogel JP, Jung J, Lavin T, Simpson G, Kluwgant D, Abalos E, Diaz V, Downe S, Filippi V, Gallos I, Galadanci H, Katageri G, Homer CSE, Hofmeyr GJ, Liabsuetrakul T, Morhason-Bello IO, Osoti A, Souza JP, Thakar R, Thangaratinam S, Oladapo OT. Neglected medium-term and long-term consequences of labour and childbirth: a systematic analysis of the burden, recommended practices, and a way forward. Lancet Glob Health. 2024 Feb;12(2):e317-e330. doi: 10.1016/S2214-109X(23)00454-0. Epub 2023 Dec 6. PMID 38070535
- [Background] Arslan, S., Okcu, G., Coşkun, A., & Temiz, F. (2019). Women'sperceptıon